CLINICAL TRIAL: NCT06244511
Title: When to Start Bipedal Exercises in Chronic Ankle Instability?
Brief Title: Bipedal vs. Unipedal Exercises in Chronic Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bezmialem Vakif University (Other); Acıbadem Atunizade Hospital (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AESKA34893209
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Instability; Ankle (Ligaments) (Old Injury)
Keywords: Proprioseptive exercise; Resistive exercise; Chronic ankle instability; Rehabilitation

STUDY DESIGN:
Intervention Model Description: There will be an equal number of participants in the two groups randomized by the computer.
Who Masked: Outcomes Assessor
Masking Description: The assessor will not know which participant received which intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Bipedal Exercise (Active Comparator): Individuals with a diagnosis of chronic ankle instability who underwent supervised exercise under the guidance of a physiotherapist for 8 weeks, 2 days a week.
  Interventions: Other: Early Bipedal Exercise
- Late Bipedal Exercise (Active Comparator): Individuals with a diagnosis of chronic ankle instability who underwent supervised exercise under the guidance of a physiotherapist for 8 weeks, 2 days a week.
  Interventions: Other: Late Bipedal Exercise

INTERVENTIONS:
Other: Early Bipedal Exercise — Proprioceptive, resistive, nuromuscular exercises and stretching; Exercise interventions involving the active use of both extremities will be implemented for the first four weeks.
  Arms: Early Bipedal Exercise
Other: Late Bipedal Exercise — Proprioceptive, resistive, nuromuscular exercises and stretching; Exercise interventions involving the active use of both extremities will be implemented for the last four weeks.
  Arms: Late Bipedal Exercise

SUMMARY:
Ankle sprain is a commonly encountered condition in clinical practice, constituting approximately 15-30% of all musculoskeletal injuries. Long-term studies have demonstrated that up to 73% of patients experience at least one more ankle sprain following an acute ankle sprain. Inadequate treatment of acute ankle instability can lead to chronic ankle instability (CAI) in 30-70% of cases.

Treatment approaches for CAI are classified into conservative and surgical methods. Typically, conservative treatment is initially employed to address proprioceptive deficits and static impairments. Passive, unidirectional treatments such as injections, electrotherapy, and ice, which do not target muscle strength, kinetic chain, tendon capacity, and cortical control, are reported to be insufficient or ineffective in treating CAI, relying solely on symptomatic relief. Therefore, therapeutic exercises are fundamental in CAI treatment, leading to positive developments in parameters such as strength, dynamic balance, functional status, quality of life, and injury risk. Among the most commonly used exercise approaches are proprioceptive and resistive exercises.

Upon reviewing the literature, it is observed that bipedal exercises have been employed from the early stages of CAI. However, due to clinical symptoms such as pain, insecurity, and fear associated with loading the affected limb, patients tend to avoid putting weight on the affected limb, resulting in the frequent use of bipedal exercises in the early phases of rehabilitation.

The aim of this study is to comparatively examine the effectiveness of unipedal exercise interventions used in the early stages of rehabilitation for individuals with CAI in terms of pain, functional stability, fear avoidance, disease severity, functional performance, balance, and patient satisfaction, in comparison to bipedal exercise interventions.

DETAILED DESCRIPTION:
Voluntary participants who have been diagnosed with chronic ankle instability will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. The study groups will be as follows: a) early bipedal exercise group, b) late bipedal exercise group.

ELIGIBILITY:
Inclusion Criteria:

* The documented unilateral ankle instability confirmed through clinical examinations (drawer test, talar tilt test) and MRI in cases requiring differential diagnosis.
* A history of an initial ankle sprain occurring at least 6 months ago.
* The presence of a recurrent sense of giving way that started at least 6 months ago and has been intermittently persistent.

Exclusion Criteria:

* Presence of a history of previous surgery in the lower extremity.
* Identification of organic and non-organic lesions such as cartilage injuries, periarticular tendon tears, and impingement syndromes.
* The existence of a fracture accompanying instability in the foot-ankle.
* Presence of congenital deformities in the foot-ankle.
* Diagnosis of talus osteochondral lesion.
* Diagnosis of ankle arthritis.
* Presence of medial ligament lesion.
* Existence of peripheral neuropathy.
* Presence of additional rheumatological diseases.
* Regular moderate-level exercise for at least 3 days a week in the last 6 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | change from baseline at 6 months
  Patients will be asked to use a 100 mm scale to indicate the intensity of ankle pain by marking a point on the scale. As the marked point approaches 100, it will represent an increase in perceived pain intensity. The location marked on the scale closer to 100 will indicate a higher level of perceived pain.
Single Leg Hop Test | 3 times for 24 weeks
  It is an athletic performance test designed to assess the functional stability of patients. In this test, participants are instructed to perform lateral hops as far as possible, and the recorded distance of their jumps serves as a score, reflecting their functional stability.
Tampa Kinesiophoby Scoring | 3 times for 24 weeks
  It is a 17-item scale developed to assess the fear of movement/re-injury.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool | 3 times for 24 weeks
  It is a 30-point, 9-item scale measuring the severity of functional ankle instability. Lower scores indicate functional ankle instability. The Minimal Clinically Important Difference for this valid and reliable scale is 3 points.
Joint Range of Motion Evaluation | 3 times for 24 weeks
  During the assessments, three repeat measurements will be made using an electronic goniometer. For goniometric measurement, the pivot point will be placed on the lateral malleolus. The fixed arm will be kept parallel to the lateral midline of the fibula. The moving arm, on the other hand, will follow the lateral midline of the 5th metatarsal bone.
Foot and Ankle Ability Measure | 3 times for 24 weeks
  This tool has been developed as a self-report instrument to comprehensively assess physical performance among individuals with various lower extremity musculoskeletal disorders, including leg, foot, and ankle conditions. It consists of 23 questions covering sub-parameters such as activity limitation, disability, and pain. Higher scores on the tool indicate greater impairment and lower function.
Star Excursion Test | 3 times for 24 weeks
  Physical performance that requires strength, flexibility, and proprioception is assessed through a dynamic test evaluating dynamic postural control and lower extremity injury risk associated with musculoskeletal injuries. The protocol of the test involves maintaining balance on the ipsilateral leg while reaching as far as possible with the contralateral leg.
Single Leg Stance Test | 3 times for 24 weeks
  Participants' standing balance will be assessed. Initially, one foot will be positioned on a firm and flat surface with the entire lower extremity in full extension, while the other lower extremity is positioned with the hip and knee flexed at 90 degrees. With their eyes closed, participants will start the timing when the foot not being tested loses contact with the ground, and the timing will stop when they place their foot back on the ground or when there is a significant increase in body sway.
Global Rating of Change Scale-GRC | 2 times for 24 weeks
  It will be used to evaluate patient satisfaction. It is designed to determine the amount of improvement or worsening of the patient over time.
  In our study, GRC consisting of 5 levels between -2 and +2 value ranges (-2: I am much worse, -1: I am worse, 0: I am the same, 1: I am better, 2: I am much better) was preferred.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Erekdağ, MSc, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Acibadem Mehmet Ali Aydinlar University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Xue X, Ma T, Li Q, Song Y, Hua Y. Chronic ankle instability is associated with proprioception deficits: A systematic review and meta-analysis. J Sport Health Sci. 2021 Mar;10(2):182-191. doi: 10.1016/j.jshs.2020.09.014. Epub 2020 Oct 2. PMID 33017672
- [Background] van den Bekerom MP, Kerkhoffs GM, McCollum GA, Calder JD, van Dijk CN. Management of acute lateral ankle ligament injury in the athlete. Knee Surg Sports Traumatol Arthrosc. 2013 Jun;21(6):1390-5. doi: 10.1007/s00167-012-2252-7. Epub 2012 Oct 30. PMID 23108678
- [Background] Hertel J. Functional Anatomy, Pathomechanics, and Pathophysiology of Lateral Ankle Instability. J Athl Train. 2002 Dec;37(4):364-375. PMID 12937557
- [Background] Malliaropoulos N, Bikos G, Meke M, Vasileios K, Valle X, Lohrer H, Maffulli N, Padhiar N. Higher frequency of hamstring injuries in elite track and field athletes who had a previous injury to the ankle - a 17 years observational cohort study. J Foot Ankle Res. 2018 Feb 26;11:7. doi: 10.1186/s13047-018-0247-4. eCollection 2018. PMID 29492109
- [Background] Diamond JE. Rehabilitation of ankle sprains. Clin Sports Med. 1989 Oct;8(4):877-91. PMID 2688911
- [Background] Dhillon MS, Patel S, Baburaj V. Ankle Sprain and Chronic Lateral Ankle Instability: Optimizing Conservative Treatment. Foot Ankle Clin. 2023 Jun;28(2):297-307. doi: 10.1016/j.fcl.2022.12.006. Epub 2023 Feb 26. PMID 37137624
- [Background] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963
- [Background] Roy A, Gupta JK, Lahiri SC. Studies on anti-inflammatory, analgesic and antipyretic activities of some indan acids. Indian J Physiol Pharmacol. 1980 Oct-Dec;24(4):310-6. PMID 6971256
- [Background] Ajis A, Maffulli N. Conservative management of chronic ankle instability. Foot Ankle Clin. 2006 Sep;11(3):531-7. doi: 10.1016/j.fcl.2006.07.004. PMID 16971246
- [Background] Martin RL, Davenport TE, Fraser JJ, Sawdon-Bea J, Carcia CR, Carroll LA, Kivlan BR, Carreira D. Ankle Stability and Movement Coordination Impairments: Lateral Ankle Ligament Sprains Revision 2021. J Orthop Sports Phys Ther. 2021 Apr;51(4):CPG1-CPG80. doi: 10.2519/jospt.2021.0302. PMID 33789434